CLINICAL TRIAL: NCT01625403
Title: Effect of Recombinant BNP on Heart and Renal Function in Acute Decompensated Heart Failure Patients With Acute Renal Injury
Brief Title: Recombinant BNP on Heart and Renal Function in Acute Heart Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Dr. Fang Yuan, Dr., Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCHESTCCU01
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Acute Heart Failure; Acute Renal Failure
Keywords: Recombinant BNP; Diuretics; Acute decompensated heart failure; Acute renal injury; Heart function; Renal function
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhBNP treated (Experimental): standard of care with rhBNP
  Interventions: Drug: rhBNP
- standard of care (Active Comparator): standard of care
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: rhBNP — intravenous administration of rhBNP 0.01 µg/kg/min
  Arms: rhBNP treated
Drug: standard of care — standard of care for heart failure
  Arms: standard of care

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant human B-type natriuretic peptide (rhBNP) on heart and renal function in patients with acute decompensated heart failure (ADHF) and acute renal injury (AKI).

DETAILED DESCRIPTION:
Patients with acute decompensated heart failure (ADHF) and acute renal injury (AKI) will be randomized to receive standard of care with or without additional rhBNP.

Clinical heart function, LVEF, SCr, GFR and other laboratory parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* acute heart failure with acute renal injury

Exclusion Criteria:

* not tolerate to rhBNP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
left ventricular systolic function | 90 days

SECONDARY OUTCOMES:
serum creatinine | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yuan, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China